CLINICAL TRIAL: NCT04197986
Title: Phase 3, Multicenter, Double-Blind, Randomized, Placebo-Controlled Trial of Infigratinib for the Adjuvant Treatment of Subjects With Invasive Urothelial Carcinoma With Susceptible FGFR3 Genetic Alterations (PROOF 302)
Brief Title: Oral Infigratinib for the Adjuvant Treatment of Subjects With Invasive Urothelial Carcinoma With Susceptible FGFR3 Genetic Alterations
Acronym: PROOF302
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The sponsor has decided to close the study due to the discontinuation of infigratinib development. The discontinuation of the study was not due to safety reasons.
Sponsor: QED Therapeutics, a BridgeBio company (Industry)
Collaborators: Helsinn Healthcare SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: QBGJ398-302; 2019-003248-63 (EudraCT Number)
Record Dates: First submitted 2019-12-02; First posted 2019-12-13 (Actual); Results first posted 2024-03-13 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-02

CONDITIONS: Upper Tract Urothelial Carcinomas; Urothelial Bladder Cancer
Keywords: FGFR3 Genetic Alterations; Upper Tract Urothelial Carcinomas; UTUC; Muscle Invasive Urothelial Carcinoma; Fibroblast Growth Factor Receptor Inhibitor; BGJ398; FGFR3; Urothelial Bladder Cancer; UBC; Infigratinib Phosphate; Infigratinib; Adjuvant; Nephroureterectomy; Distal ureterectomy; Cystectomy
MeSH Terms: interventions — infigratinib; Drug Evaluation

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned (1:1) to receive oral infigratinib phosphate or placebo
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: As a double-blind study, participants, investigators, study monitor(s) and the clinical study team will be blinded to the treatment administered.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Infigratinib 125 mg (Experimental): Participants will be randomly assigned (1:1) to receive oral infigratinib administered once daily for the first 3 weeks (21 days) of each 28-day cycle for a maximum of 52 weeks
  Interventions: Drug: Infigratinib
- Placebo (Placebo Comparator): Participants will be randomly assigned (1:1) to receive oral placebo administered once daily for the first 3 weeks (21 days) of each 28-day cycle for a maximum of 52 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Infigratinib — Participants randomly assigned to infigratinib will receive hard gelatin capsules for oral administration of infigratinib 125 mg once a day (administered as one 100-mg capsule and one 25-mg capsule) using a 3 weeks on (Days 1-21) /1 week off (Days 22-28) dosing schedule.
  Other Names: IP; Study drug
  Arms: Infigratinib 125 mg
Drug: Placebo — Participants randomly assigned to placebo will receive placebo matching in appearance the investigational product (infigratinib), which will be provided as hard gelatin capsules for oral use and will be administered once daily on a 3 weeks on (Days 1-21) /1 week off (Days 22-28) dosing schedule.
  Arms: Placebo

SUMMARY:
This is a Phase 3 multicenter, double-blind, randomized, placebo-controlled study to evaluate the efficacy of infigratinib (an oral targeted FGFR1-3 inhibitor) versus placebo, as adjuvant treatment following surgery in adult subjects with invasive urothelial carcinoma and susceptible FGFR3 genetic alterations (mutations, and gene fusions or rearrangements) who have disease that is considered at high risk for recurrence with surgery alone. The study enrolls subjects with either bladder cancer post radical cystectomy or upper tract urothelial cancer post distal ureterectomy and/or nephrectomy. Study treatment is randomized 1:1 between infigratinib or placebo with treatment up to 1 year or until invasive local, distal, or metastatic disease recurrence confirmed by independent imaging reviewer.

ELIGIBILITY:
Key Inclusion Criteria

1. Are randomized within 120 days following nephroureterectomy, distal ureterectomy or cystectomy.
2. Have histologically or cytologically confirmed, invasive urothelial carcinoma with susceptible FGFR3 alterations. Variant histology is allowed provided urothelial carcinoma is predominant (>50%). Neuroendocrine (including small and large cell), sarcomatoid, and plasmacytoid variants are excluded (any component).

   1. Regarding samples and documentation of FGFR3

      * i. FGFR3 mutation is confirmed if: FGFR3 gene is mutated in Exon 7 (R248C, S249C), Exon 10 (G370C, A391E, Y373C), or Exon 15 (K650M/T, K650E/Q)

      OR
      * ii. FGFR3 gene fusion or FGFR3 rearrangement is confirmed based on the following genomic criteria if:

        * Any fusion/rearrangement with a literature-derived known partner gene regardless of strand or frame.
        * Fusion/rearrangements in the same strand that are in frame with a novel partner gene.
        * Fusion/rearrangements with one breakpoint in the intron 17 - exon 18 hotspot region and the other breakpoint in an intergenic region or another gene. This rule excludes 3' duplications comprising only exon 18.
      * iii. The amino acid numbers for the FGFR3 mutations refer to the functional FGFR3 isoform 1 (NP_000133.1) that is the NCBI Refseq ID used to report genetic alterations in FGFR3 by the FoundationOne® CDx test (F1CDx, Foundation Medicine, USA).
      * iv. FGFR3 alteration must be confirmed by Foundation Medicine for F1CDx testing:

        * The tumor sample to be used should be from the definitive surgical resection (cystectomy, nephroureterectomy, or distal ureterectomy), or from an archival biopsy of confirmed invasive urothelial carcinoma (≥pT2).
   2. If status post neoadjuvant chemotherapy, pathologic stage at surgical resection must be Stage ≥ ypT2 and/or yN+. Prior neoadjuvant therapy is defined as at least 3 cycles of neoadjuvant cisplatin-based chemotherapy with a planned cisplatin dose of 70 mg/m2/cycle. Subjects who received less than this or non-cisplatin-based neoadjuvant treatment are not excluded.
   3. If not status post neoadjuvant chemotherapy, is ineligible to receive cisplatin-based adjuvant chemotherapy based on Galsky criteria:
   4. Subjects who refuse cisplatin-based chemotherapy or who are ineligible to receive cisplatin-based chemotherapy based on Galsky criteria must also meet the following criteria:
   5. Must have a centrally reviewed negative postoperative computed tomography (CT) (defined as lymph nodes with short axis <1.0 cm and without growth and no distant metastases according to [RECIST v1.1 criteria or negative biopsy within 28 days before randomization to confirm absence of disease at baseline.
3. Have Eastern Cooperative Oncology Group (ECOG) performance status of ≤2.
4. If a woman of childbearing potential, must have a negative pregnancy test within 7 days of the first dose of study drug. Sexually active males must use a condom during intercourse while taking study drug and for 1 month after the last dose of study drug and should not father a child during this period

Key Exclusion Criteria:

1. Presence of positive invasive surgical margins following nephroureterectomy, distal ureterectomy, or cystectomy. In subjects not eligible for further surgery, radiotherapy, or other efficacious treatment, microscopic positive noninvasive margins (eg, carcinoma in situ) without gross residual disease are allowed.
2. Have received Bacillus Calmette-Guerin (BCG) or other intravesical therapy for Non-Muscle Invasive Bladder Cancer (NMIBC) within the previous 30 days.
3. Are currently receiving or are planning to receive during participation in this study, treatment with agents that are known moderate or strong inducers or inhibitors of CYP3A4 and medications which increase serum phosphorus and/or calcium concentration. Prior anticancer or other therapies are restricted as follows:

   1. Prior adjuvant treatment for urothelial cancer is not allowed.
   2. Prior neoadjuvant therapy (eg, chemotherapy, immunotherapy, or investigational) is allowed if inclusion criterion #4 is met. Prior neoadjuvant chemotherapy must have been completed within a period of time that is greater than the cycle length used for that treatment before first dose of study drug.
   3. Prior biologic, immunotherapy, or investigational therapy should have been completed within a period that is ≥5 half-lives or 30 days, whichever is shorter, before the first dose of study drug.
4. Have previously or currently is receiving treatment with a mitogen-activated protein kinase (MEK) or selective FGFR inhibitor.
5. Have a history of primary malignancy within the past 3 years other than (1) invasive UBC or UTUC (ie, disease under study), (2) noninvasive urothelial carcinoma, (3) any adequately treated in situ carcinoma or non-melanoma carcinoma of the skin, (4) any other curatively treated malignancy that is not expected to require treatment for recurrence during participation in the study, or (5) an untreated cancer on active surveillance that may not affect the subject's survival status for ≥3 years based on clinician assessment/statement and with medical monitor approval.
6. Have current evidence of corneal keratopathy or retinal disorder confirmed by ophthalmic examination. Subjects with asymptomatic ophthalmic conditions assessed by the investigator to pose minimal risk for study participation may be enrolled in the study.
7. Have a history and/or current evidence of extensive tissue calcification
8. Have impaired gastrointestinal (GI) function or GI disease that may significantly alter the absorption of oral infigratinib
9. Have current evidence of endocrine alterations of calcium/phosphate homeostasis (eg, parathyroid disorders, history of parathyroidectomy, tumor lysis, tumoral calcinosis), unless well controlled.
10. Have consumed grapefruit, grapefruit juice, grapefruit hybrids, pomegranates, star fruits, pomelos, or Seville oranges or products containing juice of these fruits within 7 days before the first dose of study drug; have taken any Chinese herbal medicine or Chinese patent medicine treatments with anticancer activity within 14 days of the first dose of study drug.
11. Have insufficient bone marrow function:

    1. Absolute neutrophil count (ANC) <1,000/mm3 (1.0 × 109/L).
    2. Platelets <75,000/mm3 (<75 × 109/L).
    3. Hemoglobin <8.5 g/dL; transfusion support is allowed if >1 week before randomization and hemoglobin remains stable.
12. Have insufficient hepatic and renal function:

    1. Total bilirubin >1.5 × upper limit of normal (ULN) of the testing laboratory (for subjects with documented Gilbert syndrome, direct bilirubin must be ≤1.5 × ULN and enrollment requires approval by the medical monitor).
    2. AST/SGOT and ALT/SGPT >2.5 × ULN of the testing laboratory.
    3. Serum creatinine >1.5 × ULN or a calculated or measured creatinine clearance of <30 mL/min.
13. Have amylase or lipase >2.0 × ULN.
14. Have abnormal calcium or phosphorus:

    1. Inorganic phosphorus higher than 1.02 × ULN of the testing laboratory.
    2. Total serum calcium (can be corrected) higher than 1.02 × ULN of the testing laboratory.
15. Have clinically significant cardiac disease including any of the following:

    1. New York Heart Association (NYHA) Class ≥2B; subjects with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the NYHA classification.
    2. Uncontrolled hypertension
    3. Presence of CTCAE v5.0 Grade ≥2 ventricular arrhythmias, atrial fibrillation, bradycardia, or conduction abnormality.
    4. Unstable angina pectoris or acute myocardial infarction ≤3 months before the first dose of study drug.
    5. Average QTcF >470 msec (males and females). Note: If the QTcF is >470 msec in the first ECG, a total of 3 ECGs separated by ≥5 minutes should be performed. If the average of these 3 consecutive results for QTcF is ≤470 msec, the subject meets eligibility in this regard.
    6. History of congenital long QT syndrome.
16. Have had a recent (≤3 months before the first dose of study drug) transient ischemic attack or stroke.
17. If female, are pregnant or nursing (lactating).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2020-03-11 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David van Veenhuyzen, M.B., Ch.B., M.Pharm.Med., Study Director — QED Therapeutics, a BridgeBio company
Locations (143):
- United States (47):
  - Arizona Oncology Associates, Tucson, Arizona
  - City of Hope - Duarte, Duarte, California
  - City of Hope, Duarte, California
  - Loma Linda University Faculty Medical Clinics, Loma Linda, California
  - USC Norris Comprehensive Cancer Center, Los Angeles, California
  - University of Colorado Cancer Center, Aurora, Colorado
  - The Urology Center of Colorado, Denver, Colorado
  - Georgetown University Medical Center, Washington D.C., District of Columbia
  - Urological Research Network CORP, Hialeah, Florida
  - Mayo Clinic - Jacksonville, Jacksonville, Florida
  - Lakeland Regional Health Hollis Cancer Center, Lakeland, Florida
  - Emory University, Atlanta, Georgia
  - Winship Cancer Institute of Emory University, Atlanta, Georgia
  - Northwestern University Feinberg School of Medicine, Chicago, Illinois
  - UChicago Medicine Duchossois Center for Advanced Medicine (DCAM) - Hyde Park, Chicago, Illinois
  - DuPage Medical Group - Warrenville Road, Lisle, Illinois
  - Indiana University Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Tulane University/Southeastern Louisiana VA Health Care, New Orleans, Louisiana
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Saint Louis University- SLUCare Academic Pavilion, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - John Theurer Cancer Center at Hackensack University Medical Center, Hackensack, New Jersey
  - New Jersey Urology - Saddle Brook, Saddle Brook, New Jersey
  - New Jersey Urology, Voorhees Township, New Jersey
  - Albany Medical Center - Division of Urology, Albany, New York
  - Associated Medical Professionals - Syracuse, Syracuse, New York
  - Duke University Cancer Center, Durham, North Carolina
  - Accellacare-DuPage Medical Group, Raleigh, North Carolina
  - Wake Forest Baptist Health, Winston-Salem, North Carolina
  - University of Toledo, Arlington, Ohio
  - Oncology Hematology Care, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - The Ohio State University College of Medicine, Columbus, Ohio
  - The University of Toledo Medical Center, Toledo, Ohio
  - Stephenson Cancer Center, Oklahoma City, Oklahoma
  - Medical University of South Carolina, Charleston, South Carolina
  - Urology Associates, Nashville, Tennessee
  - Harold C. Simmons Comprehensive Cancer Center, Dallas, Texas
  - Bayor College of Medicine, Houston, Texas
  - Houston Methodist Hospital- Department of Urology, Houston, Texas
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - UT Southwestern, Richardson, Texas
  - Urology San Antonio, San Antonio, Texas
  - Huntsman Cancer Institute and Hospital, Salt Lake City, Utah
  - Seattle Cancer Care Alliance, Seattle, Washington
  - West Virginia University, Morgantown, West Virginia
- Belgium (4):
  - CHU de Liège - Sart Tilman, Liège, Liège/Belgium
  - ZNA Middelheim, Antwerp
  - Cliniques Universitaires Saint-Luc, Brussels
  - Universitair Ziekenhuis Leuven, Leuven
- Bulgaria (3):
  - University Multiprofile Hospital For Active Treatment Deva Maria, Burgas
  - University Multiprofile Hospital For Active Treatment Dr. Georgi Stranski EAD, Pleven
  - Multiprofile Hospital For Active Treatment "Sveta Sofia", Sofia
- Canada (6):
  - Cross Cancer Institute, Edmonton, Alberta
  - BC Cancer- Vancouver, Vancouver, British Columbia
  - Princess Margaret Cancer Centre, Toronto, Ontario
  - McGill University Health Centre (MUHC), Montreal, Quebec
  - CHU de Québec Université Laval, Québec
  - BC Cancer - Vancouver, Vancouver
- France (15):
  - Centre de Lutte Contre le Cancer - Centre Léon Bérard, Lyon, Auvergne-Rhône-Alpes
  - CHU de Nantes Hopital Hotel Dieu, Paris, Paris/France
  - Institut de Cancerologie Strasbourg Europe, Strasbourg, Strasbourg/France
  - Institut Claudius Regaud, Toulouse, Toulouse/France
  - Gustave Roussy, Villejuif, Villejuif/France
  - Hôpital Morvan, Brest
  - CHU de Nantes Hopital Hotel Dieu, Nantes
  - Hopital Bichat - Claude - Bernard, Paris
  - Centre Eugène Marquis, Rennes
  - Centre Hospitalier Privé Saint-Grégoire, Saint-Grégoire
  - Institut De Cancerologie De L'ouest - Site Saint-Herblain, Saint-Herblain
  - Clinique Mutualiste de l'Estuaire, Saint-Nazaire
  - Gustave Roussy, Villejuif
  - Hôpital Universitaire Pitié Salpêtrière, Paris, Île-de-France Region
  - Hôpital Européen Georges-Pompidou, Paris, Île-de-France Region
- Germany (13):
  - Charité - Universitatsmedizin Berlin, Berlin, Berlin/Germany
  - Urologicum Duisburg, Duisburg, North Rhine-Westphalia
  - Universitätsklinikum Düsseldorf, Düsseldorf, North Rhine-Westphalia
  - Universitätsklinikum Essen, Essen, North Rhine-Westphalia
  - Marien Hospital Herne - Universitätsklinikum der Ruhr-Universität Bochum, Herne, North Rhine-Westphalia
  - Charite Universitaetsmedizin Berlin, Berlin
  - Urologie, Berlin
  - University Hospital Duesseldorf, Düsseldorf
  - Universitätsklinikum des Saarlandes Klinik für Urologie & Kinderurologie, Homburg
  - Universitatsklinikum des Saarlandes Klinik fur Urologie & Kinderurologie, Homburg/saar
  - Universitatsklinikum Magdeburg, Magdeburg
  - Caritas-Krankenhaus St. Josef Klinik für Urologie, Regensburg
  - Universitätsklinikum Tübingen, Tübingen
- Greece (3):
  - Henry Dunant Hospital Center, Athens, Attica
  - Bioclinic Thessalonikis, Thessaloniki, Makedonia
  - Anassa General Clinic, Volos
- Italy (27):
  - Ospedale di Cremona, Cremona, Cremona/Italy
  - Ospedale Policlinico San Martino, Genova, Genova/Italy
  - Istituto Scientifico Romagnolo per lo Studio e la Cura dei Tumori, Meldola, Meldola/Italy
  - Istituto Europeo di Oncologia, Milan, Milano/Italy
  - Istituto Nazionale Tumori IRCCS Fondazione G. Pascale, Napoli, Naples
  - Azienda Ospedaliero-Universitaria Pisana, Pisa, Pisa/italy
  - IRCCS Centro di Riferimento Oncologico di Basilicata, Rionero in Vulture, Potenza
  - Arcispedale Santa Maria Nuova, Reggio Emilia, Reggio Emilia/Italy
  - Università Campus Bio-Medico di Roma, Roma, Roma/Italy
  - Azienda Ospedaliero - Universitaria San Luigi Gonzaga, Orbassano, Torino
  - Ospedale di Trento - Presidio Ospedaliero Santa Chiara, Trento, Trentino-Alto Adige
  - Centro di Riferimento Oncologico, Aviano
  - Azienda Universitaria Ospedaliera Consorziale - Policlinico di Bari, Bari
  - A.O.U.C. Polclinico di Bari U.O. Oncologia Medica Universitaria, Bari
  - ASST Cremona, Casalmaggiore
  - Ospedale Policlinico San Martino Irccs, Genova
  - Istituto Scientifico Romagnolo per lo Studio e la Cura dei Tumori, Meldola
  - Fondazione IRCCS INT Milano, Milan
  - Istituto Europeo di Oncologia, Milan
  - Int Pascale Napoli, Napoli
  - AOU San Luigi Gonzaga, Orbassano
  - Azienda Ospedaliero-Universitaria Pisana, Pisa
  - IRCCS di Reggio Emilia, Reggio Emilia
  - Policlinico Universitario Campus Biomedico, Roma
  - Citta Della Salute e Della Scienz - Torino, Torino
  - Ospedale di Trento - Presidio Ospedaliero Santa Chiara, Trento
  - IRCCS Centro di Riferimento Oncologico di Basilicata, Volterra
- Netherlands (3):
  - Canisius-Wilhelmina Ziekenhuis, Nijmegen, Gelderland
  - The Netherlands Cancer Institute, Amsterdam
  - Zuyderland MC locatie Sittard, Geleen
- Spain (20):
  - VHIO, Barcelona, Barcelona/Spain
  - Sofia, Barcelona, Barcelona/Spain
  - Institut Català d'Oncologia - Hospital Duran i Reynals (ICO L'Hospitalet), Barcelona, Barcelona/Spain
  - Institut Català d'Oncologia Badalona, Badalona, Barcelona
  - Hospital Parc Taulí de Sabadell, Sabadell, Barcelona
  - Hospital Universitario Reina Sofía, Córdoba, Córdoba/Spain
  - Institut Català d'Oncologia Girona, Girona, Girona/Spain
  - Hospital Universitario Puerta Hierro-Majadahonda, Majadahonda, Madrid
  - MD Anderson Cancer Center Madrid, Madrid, Madrid/Spain
  - Hospital Universitario Ramon y Cajal, Madrid, Madrid/Spain
  - Hospital Clinico San Carlos, Madrid, Madrid/Spain
  - Hospital Universitario 12 de Octubre, Madrid, Madrid/Spain
  - Hospital Universitario La Paz, Madrid, Madrid/Spain
  - Hospital Universitario HM Sanchinarro, Madrid, Madrid/Spain
  - Hospital Universitario Virgen del Rocio, Seville, Sevilla/Spain
  - Hospital Virgen De La Salud, Toledo, Toledo/Spain
  - Fundacion Instituto Valenciano de Oncologia, Valencia, València
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital del Mar, Barcelona
  - Althaia Xarxa Assistencial Universitària de Manresa, Manresa
- United Kingdom (2):
  - Guy's and St Thomas' NHS Foundation Trust, London
  - Lister Hospital, Stevenage

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Szymaniak J, Porten SP. Which Biomarkers are Useful in the Management of Muscle-invasive Bladder Cancer in 2022? Eur Urol Focus. 2022 Jul;8(4):901-903. doi: 10.1016/j.euf.2022.08.009. Epub 2022 Sep 2. PMID 36058810
- [Derived] Pal SK, Somford DM, Grivas P, Sridhar SS, Gupta S, Bellmunt J, Sonpavde G, Fleming MT, Lerner SP, Loriot Y, Hoffman-Censits J, Valderrama BP, Andresen C, Schnabel MJ, Cole S, Daneshmand S. Targeting FGFR3 alterations with adjuvant infigratinib in invasive urothelial carcinoma: the phase III PROOF 302 trial. Future Oncol. 2022 Jul;18(21):2599-2614. doi: 10.2217/fon-2021-1629. Epub 2022 May 24. PMID 35608106

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with a diagnosis of invasive urothelial carcinoma were recruited to this double-blind, randomized, placebo-controlled global study across 30 study centers (11 in North America, and 19 in Western Europe) based on documented evidence of FGFR3 genetic alteration. The first participant was treated on 18 March 2020. The data cutoff for the primary analysis was 28 February 2023.
Pre-assignment Details: Subjects meeting inclusion/exclusion criteria were randomly assigned 1:1 to receive oral infigratinib 125 mg (N=20) or placebo (N=19). Randomization was stratified by lymph node involvement (yes/no), prior neoadjuvant cisplatin chemotherapy (yes/no), stage (pT2 vs > pT2), and disease (upper tract urothelial carcinoma [UTUC] vs urinary bladder cancer [UBC]).
Groups:
- Infigratinib 125 mg: Participants were randomly assigned (1:1) to receive oral infigratinib administered once daily for the first 3 weeks (21 days) of each 28-day cycle for a maximum of 52 weeks.
  Infigratinib: Participants randomly assigned to infigratinib received hard gelatin capsules for oral administration of infigratinib 125 mg once a day (administered as one 100-mg capsule and one 25-mg capsule) using a 3 weeks on (Days 1-21) /1 week off (Days 22-28) dosing schedule.
- Placebo: Participants were randomly assigned (1:1) to receive oral placebo administered once daily for the first 3 weeks (21 days) of each 28-day cycle for a maximum of 52 weeks.
  Placebo: Participants randomly assigned to placebo received placebo matching in appearance the investigational product (infigratinib) provided as hard gelatin capsules for oral use and administered once daily on a 3 weeks on (Days 1-21) /1 week off (Days 22-28) dosing schedule.
Period: Overall Study
Arm/Group | Infigratinib 125 mg | Placebo
Started | 20 | 19
Treatment Ended (Per protocol, patients continued treatment for a maximum of 52 weeks (13 cycles), or until confirmed local/regional or contralateral invasive or metastatic recurrence.) | 20 | 19
Completed | 20 | 19
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Infigratinib: 125 mg oral infigratinib once daily for the first 3 weeks (21 days) of each 28-day cycle
- Placebo: Placebo once daily for the first 3 weeks (21 days) of a 28-day treatment cycle
- Total: Total of all reporting groups
Arm/Group | Infigratinib | Placebo | Total
Number analyzed (Participants) | 20 | 19 | 39
Age, Categorical [Count of Participants; unit: Participants]
  Age Group: <=18 years | 0 | 0 | 0
  Age Group: Between 18 and 65 years | 8 | 4 | 12
  Age Group: >=65 years | 12 | 15 | 27
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.1 (12.10) | 69.7 (12.75) | 67.8 (12.39)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 6
  Male | 18 | 15 | 33
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 17 | 16 | 33
  More than one race | 0 | 2 | 2
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Number; unit: participants] — North America includes United States and Canada; Europe includes Germany, Spain, France, Italy, Netherlands, and Belgium
  participants
    North America | 8 | 6 | 14
    Europe | 12 | 13 | 25
BMI [Mean (Standard Deviation); unit: kg/m2] — Population: Not available for 3 participants
  kg/m2
    number analyzed (Participants) | 19 | 17 | 36
    (all) | 27.78 (4.882) | 26.05 (4.793) | 26.96 (4.850)
ECOG PS [Count of Participants; unit: Participants] — Functional status was assessed at baseline using the Eastern Cooperative Oncology Group Performance Scale (ECOG PS), defined as follows:
  0. Fully active, able to carry out all pre-disease performance without restriction.
  1. Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature.
  2. Ambulatory and capable of all selfcare but unable to carry out any work activities; up and about more than 50% of waking hours.
  3. Capable of only limited selfcare; confined to bed or chair more than 50% of waking hours.
  4. Completely disabled.
  Participants
    0 | 15 | 11 | 26
    1 | 5 | 8 | 13
Primary Site of Cancer [Count of Participants; unit: Participants]
  UTUC | 11 | 12 | 23
  UBC | 9 | 7 | 16
Histological Subtype [Count of Participants; unit: Participants]
  Urothelial | 11 | 7 | 18
  Papillary urothelial | 7 | 8 | 15
  Mixed | 2 | 4 | 6
Screening Diagnosis Category (Pathologic Stage at Definitive Surgery) - Tumor (T) [Count of Participants; unit: Participants] — Tumor (T). T1, T2, T3, T4: Refers to the size and/or extent of the main tumor. The higher the number after the T, the larger the tumor or the more it has grown into nearby tissues.
  Participants
    T1 | 0 | 1 | 1
    T2 | 7 | 5 | 12
    T3 | 12 | 11 | 23
    T4 | 1 | 2 | 3
Screening Diagnosis Category (Pathologic Stage at Definitive Surgery) - Node (N) [Count of Participants; unit: Participants] — Node (N) refers to the number of nearby lymph nodes that have cancer. NX: Cancer in nearby lymph nodes cannot be measured; N0: There is no cancer in nearby lymph nodes; N1, N2, N3: Refers to the number and location of lymph nodes that contain cancer. The higher the number after the N, the more lymph nodes that contain cancer.
  Participants
    NX | 8 | 6 | 14
    N0 | 9 | 8 | 17
    N1 | 1 | 3 | 4
    N2 | 2 | 2 | 4
Time from Initial Diagnosis to Randomization (Days) [Mean (Standard Deviation); unit: days] | 166.2 (91.15) | 393.7 (837.30) | 277.0 (591.19)
Type of FGFR3 Alteration (Local) [Count of Participants; unit: Participants]
  Mutation | 1 | 0 | 1
  Fusion | 0 | 2 | 2
  Rearrangement | 0 | 0 | 0
  Not available | 19 | 17 | 36
FGFR3 Mutation Result (Local) [Count of Participants; unit: Participants]
  G370C | 1 | 0 | 1
  Not available | 19 | 19 | 38
FGFR3 Fusion Result (Local) [Count of Participants; unit: Participants]
  Fusion Positive - Fusion partner known | 0 | 1 | 1
  Not available | 20 | 18 | 38
Type FGFR3 Alteration (Central) [Count of Participants; unit: Participants]
  Mutation | 13 | 13 | 26
  Fusion | 6 | 4 | 10
  Rearrangement | 0 | 0 | 0
  Not available | 1 | 2 | 3
FGFR3 Mutation Result (Central) [Count of Participants; unit: Participants]
  G370C | 0 | 1 | 1
  K650E | 1 | 0 | 1
  R248C | 1 | 2 | 3
  S249C | 9 | 7 | 16
  Y373C | 2 | 3 | 5
  Not available | 7 | 6 | 13
FGFR3 Fusion Result (Central) [Count of Participants; unit: Participants]
  Y | 6 | 4 | 10
  Not available | 14 | 15 | 29
Tumor Mutational Burden [Count of Participants; unit: Participants]
  Low | 17 | 13 | 30
  High | 2 | 3 | 5
  Unknown | 0 | 2 | 2
  Cannot be determined | 0 | 1 | 1
  Not available | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Centrally Determined Disease-free Survival (DFS)
Description: DFS was defined as the number of months from date of randomization to local/regional invasive or metastatic recurrence or death due to any cause (referred as DFS event), whichever occurs earlier.
  Due to early termination of the study by the sponsor, results will focus primarily on the primary and key secondary endpoints of the study. Due to early termination of the study by the sponsor, data were censored for 85.0% to 89.5% of all subjects. Data cutoff 28 Feb 2023.
Time Frame: The number of months from date of randomization to local/regional invasive or metastatic recurrence or death due to any cause.
Population: Intent-to-treat (ITT) population, which included all subjects who were randomized
Measure: Median (Full Range); unit: Months
Groups:
- Infigratinib 125 mg: Infigratinib 125 mg once daily (3 weeks on / 1 week off treatment)
- Placebo: Placebo once daily (3 weeks on / 1 week off treatment)
Arm/Group | Infigratinib 125 mg | Placebo
Number analyzed (Participants) | 3 | 2
Months | 5.3 [0.03 to 17.48] | 5.4 [0.03 to 20.90]

2. Secondary Outcome: Investigator-assessed DFS
Description: DFS was defined as the number of months from date of randomization to local/regional invasive or metastatic recurrence or death due to any cause (referred as DFS event), whichever occurs earlier. Due to early termination of the study by the sponsor, data were censored for 85.0% to 89.5% of all subjects. Data cutoff 28 Feb 2023.
Time Frame: as for outcome 1
Population: ITT population includes all subjects who were randomized
Measure: Median (Full Range); unit: Months
Arm/Group | Infigratinib 125 mg | Placebo
Number analyzed (Participants) | 7 | 3
Months | 6.39 [0.03 to 18.07] | 12.22 [0.03 to 21.36]

3. Secondary Outcome: Metastasis-free Survival (MFS)
Description: MFS was defined as the time from randomization to any metastatic recurrence as determined by the investigator, or death due to any cause, whichever occurred earlier. Due to early termination of the study by the sponsor, data were censored for 85.0% to 89.5% of all subjects. Data cutoff 28 Feb 2023.
Time Frame: The time from randomization to any metastatic recurrence as determined by the investigator, or death due to any cause.
Population: ITT Population
Measure: Median (Full Range); unit: Months
Arm/Group | Infigratinib 125 mg | Placebo
Number analyzed (Participants) | 3 | 2
Months | 6.5 [0.03 to 18.07] | 12.2 [0.03 to 21.36]

4. Secondary Outcome: Overall Survival (OS)
Description: Overall survival time was defined as the number of months from randomization to death. Due to early termination of the study by the sponsor, data were censored for 85.0% to 89.5% of all subjects. Data cutoff 28 Feb 2023.
Time Frame: The number of months from randomization to death.
Population: ITT population
Measure: Median (Full Range); unit: Months
Arm/Group | Infigratinib 125 mg | Placebo
Number analyzed (Participants) | 20 | 19
Months | 13.1 [0.76 to 32.07] | 16.7 [1.22 to 31.57]

5. Secondary Outcome: Investigator-reviewed DFS Including Intraluminal Low-Risk Recurrence
Description: Investigator assessment of intraluminal low-risk recurrence as assessed by DFS. Due to early termination of the study by the sponsor, data were censored for 85.0% to 89.5% of all subjects. Data cutoff 28 Feb 2023.
Time Frame: as for outcome 1
Population: ITT population
Measure: Median (Full Range); unit: Months
Arm/Group | Infigratinib 125 mg | Placebo
Number analyzed (Participants) | 7 | 4
Months | 5.29 [0.03 to 18.07] | 5.62 [0.03 to 20.90]

6. Secondary Outcome: Number of Participants With Adverse Events (AEs)
Description: Number of participants with AEs
Time Frame: From first dose to last dose of study treatment +30 days (an average of 4 months for the infigratinib arm and 8 months for the placebo arm).
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Infigratinib 125 mg | Placebo
Number analyzed (Participants) | 20 | 19
Participants | 19 | 16

7. Secondary Outcome: Number of Participants With Serious Adverse Events (SAEs)
Description: Number of Participants with SAEs
Time Frame: as for outcome 6
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Infigratinib 125 mg | Placebo
Number analyzed (Participants) | 20 | 19
Participants | 2 | 2

ADVERSE EVENTS:
Time Frame: From first administration of study treatment and up to last administration of study treatment + 30 days (an average of 4 months for the infigratinib arm and 8 months for the placebo arm).
Description: AEs were assessed by the investigator according to the CTCAE version 5.0 and coded using MedDRA version 23.1.
  Treatment-emergent AEs are reported and include all AEs with onset after the first administration of study treatment and up to last administration of study treatment + 30 days if subjects ended study treatment. For a subject who had not ended study treatment, all the AEs after the first administration of study drug were considered treatment-emergent.
Arm/Group | Infigratinib 125 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 2/20 | 1/19
Serious Adverse Events (participants affected / at risk) | 2/20 | 2/19
Other Adverse Events (participants affected / at risk) | 19/20 | 16/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Infigratinib 125 mg (N=20) | Placebo (N=19)
Diarrhoea (Gastrointestinal disorders) | 2 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Urosepsis (Infections and infestations) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Chronic kidney disease (Renal and urinary disorders) | 1 | 0
Urinary tract obstruction (Renal and urinary disorders) | 0 | 1
Lymphocele (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Infigratinib 125 mg (N=20) | Placebo (N=19)
Vision blurred (Eye disorders) | 3 | 2
Diarrhoea (Gastrointestinal disorders) | 12 | 2
Dry mouth (Gastrointestinal disorders) | 7 | 1
Abdominal pain (Gastrointestinal disorders) | 3 | 1
Constipation (Gastrointestinal disorders) | 3 | 1
Nausea (Gastrointestinal disorders) | 2 | 2
Fatigue (General disorders) | 6 | 3
Mucosal inflammation (General disorders) | 4 | 2
COVID-19 (Infections and infestations) | 0 | 5
Urinary tract infection (Infections and infestations) | 1 | 3
Blood creatinine increased (Investigations) | 9 | 3
Lipase increased (Investigations) | 4 | 1
Hyperphosphataemia (Metabolism and nutrition disorders) | 12 | 0
Decreased appetite (Metabolism and nutrition disorders) | 4 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 3
Dysgeusia (Nervous system disorders) | 5 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 8 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 3 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-05-19): https://cdn.clinicaltrials.gov/large-docs/86/NCT04197986/Prot_000.pdf
  • Statistical Analysis Plan (2023-02-24): https://cdn.clinicaltrials.gov/large-docs/86/NCT04197986/SAP_001.pdf